CLINICAL TRIAL: NCT06930378
Title: Sensory Restoration in DIEP Free Flaps for Post-Mastectomy Breast Reconstruction After Breast Cancer: Comparing Non-sensitized Standard Technique to Direct Nerve Suture and to Autograft: A Three-arm, Randomized, Double-blinded Superiority Trial
Brief Title: Improvement in Breast Skin Sensibility After Breast Reconstruction: a Comparison of 3 Surgical Techniques
Acronym: S-DIEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia Esther Engels (Other)
Responsible Party: Sponsor-Investigator, Patricia Esther Engels, Principal Investigator, Consultant and Senior Clinical Researcher, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNCTP000006257; BASEC2024-02109 (Other: BASEC (Business Administration System for Ethics Committees) Switzerland)
Record Dates: First submitted 2025-03-03; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Surgery; Reconstruction Breast Surgery; Sensitization; DIEP Flap Breast Reconstruction
Keywords: free flap; breast reconstruction; autologous-based reconstruction; neurotization; sensory recovery; post-mastectomy sensation; autologous breast reconstruction; DIEP flap

STUDY DESIGN:
Intervention Model Description: Three-arm, Randomised, Double-blinded Superiority Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- no nerve suture (No Intervention): No nerve suture will be carried out.
- direct nerve suture (Experimental): Epineural coaptation of one nerve of the flap to one nerve of the breast region
  Interventions: Procedure: Nerve Suture
- interposition of an autograft (Experimental): Epineural coaptation intercostal nerve flap to autograft (from another intercostal nerve of the flap) to intercostal nerve of the breast = interposition of an autograft
  Interventions: Procedure: Nerve Suture

INTERVENTIONS:
Procedure: Nerve Suture — Sensory nerve coaptations will be performed
  1. either by suturing the donor to the recipient nerve immediately (1 coaptation)
  2. or by interposing an autograft originating from the zone of the flap to be discarded (2 coaptations). The anterior cutaneous branch (ACB) of the 3rd or 4th intercostal nerve (ICN) will be connected to the sensory branch of the 10th, 11th or 12th ICN of the flap.
  Arms: direct nerve suture; interposition of an autograft

SUMMARY:
The goal of this clinical trial is to learn if nerve sutures in free flap breast reconstruction can optimize sensibility in the reconstructed breast in patients opting for DIEP flap breast reconstruction due to breast cancer or genetic conditions. Affected women 18 to 80 years old can be included. The main question is:

If a nerve suture was carried out, can pressure be felt better on the reconstructed breast after 12 months? If a nerve suture was carried out, will better sensibility and quality of life be felt and perceived (questionnaire) at 12 and 24 months after the initial operation ? Researchers will compare two different nerve suture techniques and no nerve suture to one another to see if and which nerve suture optimizes sensibility.

Participants will have regular visits and follow-up controls, during which

* their sensibility will be tested multimodally,
* they will fill out questionnaires
* skin biopsies will be taken.

DETAILED DESCRIPTION:
Breast reconstruction with autologous tissue is one of the most important methods: The DIEP (deep inferior epigastric artery perforator) flap is today's workhorse in autologous reconstruction. Routinely, the arteries and veins of the donor- and recipient sites are connected, but not the nerves. The sensory recovery is an undervalued aspect despite the disadvantages of insensate flaps. Connection of the abdominal flap skin's nerves to the breast region's nerves allows sensitized reconstruction. The research project aims to make sensitized flap-based breast reconstruction the standard method by proving its superiority, using the sensory testing with Semmes-Weinstein-Monofilament (pressure threshold) as the primary outcome measured before surgery and 12 months post-surgery. Therefore, patients will be randomized in three groups:

1. sensitization with direct nerve suture or
2. autograft or
3. no sensitization. Moreover, no previous studies have analyzed the potential changes in flap skin with proteomics, thus justifying our secondary objective.

The hypothesis is that flaps with nerve suture(s) have better sensibility. The main outcome will be the sensory testing (pressure threshold). As secondary outcomes the questionnaire will show the patients' quality of life, and the proteomic analysis, should, according to our hypothesis, show that quantity and expression of the proteins of flap skin with nerve suture are closer to normal skin than without nerve suture.

ELIGIBILITY:
A) Pilot study

Inclusion criteria:

* 18-80 years old
* having received DIEP flap breast reconstruction with a flap not completely buried
* having given written informed consent for participating in the study

Exclusion criteria:

* postoperative radiotherapy on the flap
* neurological conditions as diabetic neuropathy, alcoholism or any other severe underlying peripheral neuropathy including chemotherapy-induced neuropathy or neuropathy induced by other medications
* active smoking
* language barrier
* pregnancy or lactating women

B) Main study

Inclusion Criteria:

* 18 to 80 years old
* having given written informed consent for participating in the study
* receiving immediate or delayed unilateral DIEP breast reconstruction with a DIEP flap which will not be completely buried

Exclusion Criteria:

* autologous reconstruction where the flap is completely buried
* patients in need of both-sided reconstruction (double DIEP)
* postoperative radiotherapy on the flap
* neurological conditions as diabetic neuropathy, alcoholism, or any other severe underlying peripheral neuropathy including chemotherapy-induced neuropathy or neuropathy induced by other medications
* active smoking
* language barrier
* pregnancy at time of planned DIEP flap surgery and lactation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — XX chromosome patients willing to have autologous breast reconstruction
Enrollment: 63 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Semmes-Weinstein-Monofilament-Test | At 12-months-follow-up
  The results of one modality of the sensory testing, the Semmes-Weinstein-Monofilament-Test for pressure perception.
  The breast will be divided into 9 zones, which will all be measured with the Semmes Weinstein monofilament 20-piece full kit (unit: grams of force) at the given time (see time frame).

SECONDARY OUTCOMES:
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  Semmes-Weinstein monoflament The breast will be divided into 9 zones, which will all be measured with the Semmes Weinstein monofilament 20-piece full kit at the given times (see time frame).
  The resulting monofilament values (unit: grams of force) are examined over the various specified periods and the delta is determined.
Sensory recovery to DIEP flap | 12 months postop
  2-point-discrimination, i.e. threshold distance between two points that are perceived as separate in millimeters. Instrument: Aesthesiometer. 9 zones of the breast.
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  2-point-discrimination, i.e. threshold distance between two points that are perceived as separate in millimeters. Instrument: Aesthesiometer. 9 zones of the breast.
  Measurement at the specified times (see time frame), determination of the delta.
Sensory recovery to DIEP flap | 12 months postop
  Vibration perception with tuning forks of 256 and 32 Hz. Binary: yes/no on 9 zones of the breast.
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  Vibration perception with tuning forks of 256 and 32 Hz. 9 zones of the breast. Binary: yes/no Evaluation of the difference in the number of zones of the breast with perception of vibration, delta over different time points.
Sensory recovery to DIEP flap | 12 months postop
  Temperature perception. Metal rods of 6°C and 37°C. Patients have to indicate which rod feels colder that the other. Capacity of differentiation of temperature: yes/no on 9 zones of the breast.
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  Temperature perception. Metal rods of 6°C and 37°C. Patients have to indicate which rod feels colder that the other. Capacity of differentiation of temperature: yes/no on 9 zones of the breast. Testing at given time points (see time frame), Calculation of delta of number of zones with distinction.
Sensory recovery to DIEP flap | 12 months postop
  Temperature surface. FLIR thermal camera, flap monitor versus whole breast and contralateral breast surface temperature, difference in temperature in degree Celsius.
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  Temperature surface. FLIR thermal camera, flap monitor versus whole breast and contralateral breast surface temperature, difference in temperature in degree Celsius. Calculation of delta over given time points (see time frame)
Sensory recovery to DIEP flap | 12 months postop
  Sharp/dull:
  Instrument system used: 18G needle / cotton swab, on nine areas of the breast.
  * Each area will be tested 3 consecutive times with both objects (i.e., 6 measurements per area)
  * The distinction between prick and gentle pressure will be considered successful if the patient responds correctly 5 times out of 6 or 6 times out of 6 (distinction ability: yes/no)
Change in breast sensation | day-1/1week/3/6/12/24 months postop
  Sharp/dull:
  Instrument system used: 18G needle / cotton swab, on nine areas of the breast.
  * Each area will be tested 3 consecutive times with both objects (i.e., 6 measurements per area)
  * The distinction between prick and gentle pressure will be considered successful if the patient responds correctly 5 times out of 6 or 6 times out of 6 (distinction ability: yes/no) Delta calculation over given time points (see time frame)
Breast-specific health-related QoL | 12 months postop
  Breast-Q®
Breast-specific health-related QoL (change over time) | Day -1, 12 &24 months postop
  Breast-Q®, delta of points over time (see time frame)
Operative time | At time of 1st operation
  Minutes for nerve coaptation(s)
Changes to DIEP flap skin | A) Pilot study Postoperatively at any time of follow-up-interventions. B) Main study At time of 1st operation and at 6-months-follow-up
  Proteomics, neuroprotein quantification
Sensory recovery to DIEP flap | 12 months postop
  2-point-discrimination, i.e. threshold distance between two points that are perceived as separate in millimeters. Instrument: Aesthesiometer.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Engels, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Puonti HK, Broth TA, Soinila SO, Hallikainen HK, Jaaskelainen SK. How to Assess Sensory Recovery After Breast Reconstruction Surgery? Clin Breast Cancer. 2017 Oct;17(6):471-485. doi: 10.1016/j.clbc.2017.04.011. Epub 2017 Apr 29. PMID 28673764
- [Background] Blondeel PN, Demuynck M, Mete D, Monstrey SJ, Van Landuyt K, Matton G, Vanderstraeten GG. Sensory nerve repair in perforator flaps for autologous breast reconstruction: sensational or senseless? Br J Plast Surg. 1999 Jan;52(1):37-44. doi: 10.1054/bjps.1998.3011. PMID 10343589
- [Background] Spiegel AJ, Salazar-Reyes H, Izaddoost S, Khan FN. A novel method for neurotization of deep inferior epigastric perforator and superficial inferior epigastric artery flaps. Plast Reconstr Surg. 2009 Jan;123(1):29e-30e. doi: 10.1097/PRS.0b013e3181905564. No abstract available. PMID 19116520
- [Background] Bijkerk E, Beugels J, van Kuijk SMJ, Lataster A, van der Hulst RRWJ, Tuinder SMH. Clinical Relevance of Sensory Nerve Coaptation in DIEP Flap Breast Reconstruction Evaluated Using the BREAST-Q. Plast Reconstr Surg. 2022 Nov 1;150(5):959e-969e. doi: 10.1097/PRS.0000000000009617. Epub 2022 Aug 22. PMID 35993852
- [Background] Shiah E, Laikhter E, Comer CD, Manstein SM, Bustos VP, Bain PA, Lee BT, Lin SJ. Neurotization in Innervated Breast Reconstruction: A Systematic Review of Techniques and Outcomes. J Plast Reconstr Aesthet Surg. 2022 Sep;75(9):2890-2913. doi: 10.1016/j.bjps.2022.06.006. Epub 2022 Jun 17. PMID 35872020
- [Background] Ducic I, Yoon J, Momeni A, Ahcan U. Anatomical Considerations to Optimize Sensory Recovery in Breast Neurotization with Allograft. Plast Reconstr Surg Glob Open. 2018 Nov 7;6(11):e1985. doi: 10.1097/GOX.0000000000001985. eCollection 2018 Nov. PMID 30881792
- [Background] Spiegel AJ, Menn ZK, Eldor L, Kaufman Y, Dellon AL. Breast Reinnervation: DIEP Neurotization Using the Third Anterior Intercostal Nerve. Plast Reconstr Surg Glob Open. 2013 Dec 6;1(8):e72. doi: 10.1097/GOX.0000000000000008. eCollection 2013 Nov. PMID 25289267
- [Background] Beugels J, Cornelissen AJM, van Kuijk SMJ, Lataster A, Heuts EM, Piatkowski A, Spiegel AJ, van der Hulst RRWJ, Tuinder SMH. Sensory Recovery of the Breast following Innervated and Noninnervated DIEP Flap Breast Reconstruction. Plast Reconstr Surg. 2019 Aug;144(2):178e-188e. doi: 10.1097/PRS.0000000000005802. PMID 31348332
- [Background] Hamilton KL, Kania KE, Spiegel AJ. Post-mastectomy sensory recovery and restoration. Gland Surg. 2021 Jan;10(1):494-497. doi: 10.21037/gs.2020.03.22. PMID 33634007
- [Background] Bijkerk E, van Kuijk SMJ, Lataster A, van der Hulst RRWJ, Tuinder SMH. Breast sensibility in bilateral autologous breast reconstruction with unilateral sensory nerve coaptation. Breast Cancer Res Treat. 2020 Jun;181(3):599-610. doi: 10.1007/s10549-020-05645-y. Epub 2020 Apr 28. PMID 32346819